CLINICAL TRIAL: NCT00666042
Title: Laboratory-masked, Randomized Parallel, Comparative, Pilot Study on the Bioavailability of Vigamox in the Aqueous Humor When Administered Either as Commercially Available Eye Drops or in a Spray Form
Brief Title: Bioequivalence of Eye Drops and Spray Administration of Vigamox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Ophthalmic Pharma (Industry)
Responsible Party: Dr. Adi Michaeli/Principal Investigator, Tel Aviv Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Eye drops vs. spray; different administrations
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2009-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Vigamox delivered as spray
  Interventions: Drug: Vigamox - administration in spray form
- B (Active Comparator): Patients will receive the commercially available Vigamox drops
  Interventions: Drug: Vigamox eye drops

INTERVENTIONS:
Drug: Vigamox - administration in spray form — Vigamox will be administered in a spray form
  Arms: A
Drug: Vigamox eye drops — Vigamox eye drops
  Arms: B

SUMMARY:
The study compares the amounts of Vigamox absorbed when administered as eye drops or in a spray form. Both administrations will be prior to patients undergoing elective cataract surgery and the aqueous samples will be analyzed by a laboratory in a masked fashion. The hypothesis is that there will be no difference between the 2 modes of administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cataract surgery

Exclusion Criteria:

* Allergy to Vigamox

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalency between the 2 ways of administration | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Adi Michaeli, MD, Principal Investigator — TAMC, Tel Aviv, Israel
Locations (1):
- Dept. of Ophthalmology, TAMC, Tel Aviv, Israel